CLINICAL TRIAL: NCT04611438
Title: A Prospective Multi-Center Single-Arm Clinical Trial on Cognitive Effect of Cannabidiol (CBD-OS®) on Dravet Syndrome and Lennox-Gastaut Syndrome
Brief Title: Research on Cognitive Effect of Cannabidiol on Dravet Syndrome and Lennox-Gastaut SyndromeGastaut Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2020-0120
Record Dates: First submitted 2019-09-16; First posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Dravet Syndrome; Lennox Gastaut Syndrome
Keywords: cannabidiol; pediatric; Dravet syndrome; Lennox-Gastaut syndrome
MeSH Terms: conditions — Epilepsies, Myoclonic; Lennox Gastaut Syndrome | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Patients would be from 2 to 18 years old diagnosed with Dravet syndrome or Lennox-Gastaut syndrome, who are intractable to more than 2 antiepileptic medications. Caregivers would purchase cannabidiol and give it to the patient according to titration schedule. Patients would go through laboratory, neuropsychologic, and electroencephalographic tests before, during and after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CBD (Experimental): The patient would be on cannabidiol for 24 weeks and would go through laboratory, electroencephalography, and neuropsychological tests before, during, and after intervention.
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — Intervention schedule for each patient is as follows:
  1. Baseline Phase (2 weeks) Baseline Phase starts from the screening visit, where the patient and caregiver write permission to the trial and goes through laboratory, electroencephalography, and neuropsychological tests.
  2. Treatment Period: Titration (2 weeks) + stabilization period (10 weeks) + maintenance period (12 weeks)
     * Titration: The patient would start cannabidiol on 5mg/kg/mg for 1 week and titrate dosage up to 10mg/kg/day for second week with the caregiver monitoring the patient's tolerability
     * Stabilization: caregiver monitoring the patient's tolerability, with no change in medication dosage
     * Maintenance: no change in medication dosage

SUMMARY:
The clinical trial "A Prospective Single-Center Single-Arm Clinical Trial on Cognitive Effect of Cannabidiol (CBD-OS®) on Dravet syndrome and Lennox-Gastaut Syndrome" is a single-group phase III study done in single tertiary referral center in Seoul, Korea.

Chief investigator is Dr. Hoon-Chul Kang of Severance Hospital, Yonsei University College of Medicine. Associate investigators are Dr. Heung Dong Kim, Joon Soo Lee, Se Hee Kim, Han Som Choi, Ji Hoon Na, Dong Hwa Yang, and Hee Jung Kang, of Severance Hospital, Yonsei University College of Medicine.

The aim of the study is to evaluate the effect of cannabidiol (CBD-OS®) on cognitive functions in patients aged from 2 to 18 years old diagnosed with Dravet syndrome or Lennox-Gastaut syndrome. The duration of study is planned as one year, after patient recruitment of 6 months. The intervention period in each patient is 24 weeks, with 2 weeks of medication titration, stabilization period of 10 weeks, and maintenance period of 12 weeks. The recruitment goal of patient number is 104, considering the study power of 90 percent.

Primary outcomes are improvement of cognitive and development and improvement of seizure outcome. Secondary outcomes are improvement in behavior and quality of life.

Safety monitoring criteria are adverse event profiles and physician's and caregiver's global assessment.

Statistical analysis of outcomes is subject only to the patients who completed the 24-week medication and 2 times of tests before and after treatment of cannabidiol. Evaluation of seizure outcomes would include all patients who completed the 24-week medication and those who dropped out of the study, either by follow-up loss or discontinuation of medication due to incomplete seizure control or adverse effect of the medication.

To evaluate safety, the investigators would measure adverse events and dropout rates by percentage. The investigators would analyze overall evaluation of the caregivers and investigator. Serious adverse events would be noted after causality evaluation.

DETAILED DESCRIPTION:
Selection criteria of the patients are as below:

1. Age: 2 years old to 18 years old
2. Investigation center: Severance hospital, Yonsei University College of Medicine, Seoul, Korea
3. A) Diagnosed as Dravet syndrome by clinical manifestations and/or genetic test B) Diagnosed as Lennox-Gastaut syndrome by clinical manifestations and electroencephalography
4. The diagnosed patients by criteria 3-(1) or 3-(2) with intractable seizures after using over two antiepileptic medications
5. Patients and caregivers who agreed to participation in this trial

Exclusion criteria of the patients are as below:

1. Patients with possibility of progressive central nervous system disease other systemic disease
2. The patients who started additional antiepileptic medication during the investigation period, with exception of short-term acute treatment of seizures (e.g. benzodiazepine for rescue therapy)
3. Patients with alanine and aspartate aminotransferase and/or total bilirubin levels over 2 times of the normal range, or blood urea nitrogen and creatinine ratio over 3 times of the normal range
4. Patient with hypersensitivity or allergic reactions to cannabidiol
5. patients who are incapable of executing cognitive tests, or cases whom the investigators consider inappropriate to be enrolled in the trial Overall trial schedule for each patient is as follows:

A) Baseline Phase (2 weeks)

* Baseline Phase starts from the screening visit, where the patient and caregiver write permission to the trial and goes through laboratory, electroencephalography, and neuropsychological tests.

B) Treatment Period : Titration(2 weeks) + stabilization period (10 weeks) + maintenance period (12 weeks)

* Titration: cannabidiol titration up to 10mg/kg/day with the caregiver monitoring the patient's tolerability
* Stabilization: caregiver monitoring the patient's tolerability, with no change in medication dosage
* Maintenance: no change in medication dosage
* Statistical analysis of outcomes would be done as follows:

T-test would be done to compare each test before and after cannabidiol treatment. For multiple results along the intervention time period, repeated data analyses would be done. Continuous variables would be evaluated by repeated measures analysis of variance or generalized estimating equations. Nominal variables would be evaluation by chi-squared test or trend test.

Evaluation of seizure outcomes would include all patients who completed the 24-week medication and those who dropped out of the study, either by follow-up loss or discontinuation of medication due to incomplete seizure control or adverse effect of the medication.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 2 years old to 18 years old
2. Investigation center: Severance hospital, Yonsei University College of Medicine, Seoul, Korea
3. (1) Diagnosed as Dravet syndrome by clinical manifestations and/or genetic test (2) Diagnosed as Lennox-Gastaut syndrome by clinical manifestations and electroencephalography
4. The diagnosed patients by criteria 3-(1) or 3-(2) with intractable seizures after using over two antiepileptic medications
5. Patients and caregivers who agreed to participation in this trial

Exclusion Criteria:

1. Patients with possibility of progressive central nervous system disease other systemic disease
2. The patients who started additional antiepileptic medication during the investigation period, with exception of short-term acute treatment of seizures (e.g. benzodiazepine for rescue therapy)
3. Patients with alanine and aspartate aminotransferase and/or total bilirubin levels over 2 times of the normal range, or blood urea nitrogen and creatinine ratio over 3 times of the normal range
4. Patient with hypersensitivity or allergic reactions to cannabidiol
5. patients who are incapable of executing cognitive tests, or cases whom the investigators consider inappropriate to be enrolled in the trial

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 107 (Estimated)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
development assessment | 24 weeks
  Assessment of cognition and development would be done by Bayley Scales of Infant Development, Wechsler Preschool and Primary Scale of Intelligence, Wechsler Intelligence Scale for Children, Developmental Test of Visual-Motor Integration, and CCTT according to the patient's age and capability.
Seizure outcome | 24 weeks
  Caregivers would report seizure outcome by Caregiver Global Impression of Change in Seizure Duration or Caregiver/patient Global Impression of Change. (CGIC)

SECONDARY OUTCOMES:
Behavior assessment | 24 weeks
  Behavior would be evaluated by Child Behavior Checklist (K-CBCL)
Quality of life assessment | 24 weeks
  Tool for evaluation quality of life is Quality of Life in Childhood Epilepsy questionnaire(K-QOLCE).

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Devinsky O, Cross JH, Laux L, Marsh E, Miller I, Nabbout R, Scheffer IE, Thiele EA, Wright S; Cannabidiol in Dravet Syndrome Study Group. Trial of Cannabidiol for Drug-Resistant Seizures in the Dravet Syndrome. N Engl J Med. 2017 May 25;376(21):2011-2020. doi: 10.1056/NEJMoa1611618. PMID 28538134
- [Result] Devinsky O, Patel AD, Cross JH, Villanueva V, Wirrell EC, Privitera M, Greenwood SM, Roberts C, Checketts D, VanLandingham KE, Zuberi SM; GWPCARE3 Study Group. Effect of Cannabidiol on Drop Seizures in the Lennox-Gastaut Syndrome. N Engl J Med. 2018 May 17;378(20):1888-1897. doi: 10.1056/NEJMoa1714631. PMID 29768152